CLINICAL TRIAL: NCT04162002
Title: Effects of Restylane® Lyft Filler Injection for Hand Rejuvenation on First Impressions
Brief Title: Restylane® Lyft Filler Injection for Hand Rejuvenation on First Impressions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DeNova Research (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Steven H. Dayan, Principal Investigator, Clinical Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REST- HAN-2019
Record Dates: First submitted 2019-08-01; First posted 2019-11-13 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Hand Rejuvination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Restylane® Lyft Filler Injection (Experimental)
  Interventions: Drug: Restylane® Lyft

INTERVENTIONS:
Drug: Restylane® Lyft — Filler Injection

SUMMARY:
The purpose of this research is to determine the effects of Restylane® Lyft Filler injection into the back of the hand on first impressions.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of ages 28 and above.
2. Subjects will be required not to have had previous filler fat injections, or other cosmetic treatments to their hands within the last 12 months.
3. Subjects that understand the purpose and aspects of the study, freely sign the consent and complete the required treatment and follow up visit. -

Exclusion Criteria:

1. Males and females below age of 28.
2. Subjects who have had previous filler, fat injections, or other cosmetic treatments to their hands within the last 12 months.
3. Subjects who are pregnant or nursing.
4. Subjects with a known allergy or sensitivity to any component of the study ingredients.
5. Any history of bleeding disorders (iatrogenic or otherwise). This includes persons who have undergone therapy with thrombolytics, anticoagulants, or inhibitors of platelet aggregation in the preceding 3 weeks.
6. Anyone taking aspirin, ibuprofen, St. John's Wort, or high doses of Vitamin E supplements in the last 3 weeks.
7. Subjects with diseases, injuries, or disabilities of the hand, including those with autoimmune disease affecting the hand, hand implants, Dupuytren's contracture, history of hand tumor, vascular malformations, Raynaud's disease and patients at risk for tendon rupture.
8. Subjects that do not understand the purpose and aspects of the study, do not sign the consent and do not complete the required treatment and follow up visit will also be excluded. -

Min Age: 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
The effects of Restylane® Lyft Filler injection into the dorsal hand on first impressions. | 4 weeks
  Subjects will have a picture of their hand evaluated by third party physicians on the basis of:
  Social Skills Positive mood, gets along with others well, friendly 1-10 rating
  Academic Performance Intelligent, highly educated, received good grades in school 1-10 rating
  Dating Success Dates frequently, lacks dating anxiety 1-10 rating
  Occupational Success Good worker, competent, motivated for success, suitable as potential employee 1-10 rating
  Attractiveness Pleasing appearance 1-10 rating
  Financial Success Has achieved financial success, member of a high social class 1-10 rating
  Relationship Success Willingness to compromise, ability to maintain long term friendships 1-10 rating
  Athletic Success Excels at athletic skills, plays individual and/or team sports 1-10 rating

CONTACTS AND LOCATIONS:
Overall Officials: Steven Dayan, MD, Principal Investigator — DeNova Research
Locations (1):
- DeNova Research, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided